CLINICAL TRIAL: NCT07180368
Title: Assessment and Management of Multiple Drug Use in Elderly Chronic Disease Patients
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ky20252065-F-1
Record Dates: First submitted 2025-06-29; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease; Diabete Mellitus; Chronic Kidney Disease; Hypertension; Heart Failure; Hyperlipidemia; Obesity &Amp; Overweight; Chronic Obstructive Pulmonary Disease (COPD); Stroke
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Renal Insufficiency, Chronic; Hypertension; Heart Failure; Hyperlipidemias; Obesity; Overweight; Pulmonary Disease, Chronic Obstructive; Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to understand the impact of polypharmacy on the prognosis of elderly patients with chronic diseases. The main research question it aims to address is:

Does polypharmacy affect the prognosis of elderly patients with chronic diseases? Elderly patients with chronic diseases will be asked to complete online survey questions regarding their disease prognosis over a 2-year period.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older with at least one chronic disease

Exclusion Criteria:

* Patients without chronic diseases
* Patients refused to participate in the study
* Patients with unstable vital signs

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with chronic diseases and multiple comorbidities
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessing the current status of polypharmacy in elderly patients with chronic diseases in Shaanxi Province via cluster sampling questionnaire survey | Start from enrollment to the end of the study at 2 years.
  A cluster sampling method was used to conduct a survey on elderly patients with chronic diseases in Shaanxi Province. A questionnaire survey was conducted in different regional locations to collect detailed medication information from patients, such as the number of chronic diseases (types), the types of medications used (types), specific drug names, medication costs (yuan), and duration of medication use (months). Medication habits, such as whether the medication is prescribed by a hospital, purchased from a pharmacy, recommended by friends, or promoted through advertisements, etc. Specific items include concerns about drugs and current physical discomforts. A 5-point Likert scale was adopted, where 1 point indicates "strongly disagree" and 5 points indicate "strongly agree". After questionnaire collection, combined with Beers, STOPP/START, and Chinese elderly PIM criteria, a polypharmacy evaluation and management strategy for these patients was developed.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China